CLINICAL TRIAL: NCT05848804
Title: Linus Health Hearing Screening Clinical Study
Brief Title: Hearing Screener Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Linus Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HSCS-001
Record Dates: First submitted 2023-04-28; First posted 2023-05-08 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Hearing Screener

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective is to compare the Linus Health Hearing Screener (LHHS) to established hearing screening methods performed by a hearing specialist. We will perform an in-office speech hearing test and compare the thresholds with those measured from the iPad at a distance of 1ft with a sound pressure level (SPL) (dBA) meter

ELIGIBILITY:
Inclusion Criteria:

* All participants must be (1) Those with a range of hearing ability but not deaf; (2) 55+ years old; (3) able to use an iPad and Apple Pencil; (4) as close to their normal hearing conditions as possible: if they wear hearing aids normally they should have them during the assessment; if not, they should not wear them; (5) able to provide written informed consent in the Institutional Review Board-approved informed consent form; (6) willing and able to comply with all study procedures as outlined in the informed consent; and (7) fluent in English.

Exclusion Criteria:

* Exclusion criteria include (1) individuals who are not able to understand or willing to comply with the directions for the administration of neuropsychological tests; (2) the presence of a major psychiatric upset such as bipolar disorder; (3) present with major medical problems such as cancer or epilepsy. Study staff will review potential participants who do not have dementia and can be approached about the study.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to three US sites will be used in this study for enrollment. Participants will be recruited from the following clinics: nursing home, memory clinic, primary and/or specialty care in order to recruit subjects with a range of hearing functions.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-22 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Hearing Thresholds | 1 Year
  The objective is to compare the Linus Health Hearing Screener (LHHS) to established hearing screening methods performed by a hearing specialist. We aim to perform an in-office hearing test and compare the thresholds with those measured from the iPad at a distance of 11ft with an SPL (dBA) meter. Comparing hearing test results between the LHHS and the results of a lab grade audiogram.

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Gomes-Osman, PhD, Study Director — Linus Health
Locations (1):
- Crossover Mangement, Wake Forest, North Carolina, United States